CLINICAL TRIAL: NCT01249755
Title: International Validation of a Delirium Prediction Model for ICU Patients (PRE-DELIRIC) in ICUs; a Multicentre Trial.
Brief Title: International Validation of a Delirium Prediction Model for ICU Patients
Status: Completed | Type: Observational
Sponsor: Radboud University Medical Center (Other)
Responsible Party: Principal Investigator, Mark van den Boogaard, PhD, Radboud University Medical Center
Other Study IDs: 20110901
Record Dates: First submitted 2010-11-26; First posted 2010-11-30 (Estimated); Last update posted 2012-08-10 (Estimated); Status verified 2012-08

CONDITIONS: Delirium
MeSH Terms: conditions — Delirium

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- delirious patients: The cohort is divided in delirious and non-delirious patients

SUMMARY:
Recently our ICU research group developed and validated a delirium prediction model in the NetherlandsThis. This model has a high predictive value. We want to examine what the predictive value is in ICUs of other European countries.

DETAILED DESCRIPTION:
Delirium is a serious and common disorder in ICU patients. It is increasingly recognized that screening of ICU patients is a valuable tool for early detection and treatment of delirium, which may reduce its incidence, severity and duration. Apart from treatment of delirium, delirium prevention (pharmacological and nursing interventions)is an important issue. However, it is time consuming to take preventive measures in all ICU patients. The recently developed prediction model facilitates the conduct of preventive measures focused on high risk groups. This prediction model is developed and validated in the Netherlands. The aim of our study is to investigate the predictive value of the model in ICUs in other countries.

ELIGIBILITY:
Inclusion Criteria:

* patients 18 years or older

Exclusion Criteria:

* delirious state within the first 24hours after ICU admission
* sustained comatose during complete ICU stay
* admission duration less than twelve hours;
* serious auditory or visual disorders
* unable to understand the language of the included centre
* severely mentally disabled
* serious receptive aphasia
* or if there are missing or incomplete delirium screenings during admission to the ICU

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult patients admitted to the ICU
Sampling Method: Non-Probability Sample
Enrollment: 2000 (Actual)
Dates: Start 2011-11; Primary Completion 2012-06 (Actual); Study Completion 2012-08 (Actual)

PRIMARY OUTCOMES:
delirium | during admission at the critical care
  Delirium is defined as at minimum one positive CAM-ICU screening during the complete ICU stay

CONTACTS AND LOCATIONS:
Overall Officials: Mark van den Boogaard, MSc, Principal Investigator — Radboud University Medical Center